CLINICAL TRIAL: NCT04000776
Title: Triple-tracer Molecular Imaging Using 18F-FDG, 68Ga-PSMA and 68Ga-OCTREOTATE to Characterize Metastatic Castration-resistant Prostate Cancer (mCRPC) and Evaluate Eligibility for Radionuclide Therapies
Brief Title: 3TMPO (Triple-Tracer Strategy Against Metastatic Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Oncopole (Unknown); Canadian Cancer Society (CCS) (Other); Merck Canada Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 3TMPO
Record Dates: First submitted 2019-06-19; First posted 2019-06-27 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Radionuclide Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Bone or soft-tissues biopsies or blood samples (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FDG Positron emission tomography (PET) scan — Patients will undergo 18F-FDG and whole-body PET/CT (vertex to thighs, or to feet if known lower-limb metastases).
  The patient will be measured and weighed before the exam in order to calculate a personalized dose. An intravenous catheter will be put in place in peripheral vein to allow injection of the tracer.
Diagnostic Test: PSMA Positron emission tomography (PET) scan — Patients will sequentially undergo 68Ga-PSMA and whole-body PET/CT (vertex to thighs, or to feet if known lower-limb metastases).
Diagnostic Test: OCTREOTATE Positron emission tomography (PET) scan — In the case a patient would present at least one PSMA-negative/FDG-positive lesion, he will be referred to undertake a whole-body 68Ga-OCTREOTATE PET/CT within 10 days of the first PET/CT. The delay between this third PET scan and the last one should be minimal (not least than 18 hours, not more than 10 days).
  Images and data will be reviewed centrally within 4 days by the Imaging Corelab, which will produce a final report confirming patient's eligibility to Radioligand therapy (RLT).
Other: Optional Bone or soft-tissue biopsies — Patients presenting FDG-positive/PSMA-negative or Octreotate-positive lesions on imaging will be asked to undergo a biopsy of these lesions (optional) for research purposes. Bone or soft-tissue biopsies will be collected by an interventional radiologist according to site's standard-of-care procedure and sent to the local pathology department for preparation (formalin-fixed and paraffin-embedded); the blocks being sent to the Pathology Corelab.

SUMMARY:
Prostate cancer (PCa) is the most common solid organ cancer in North American men. Patients becoming refractory to loco-regional therapy receive androgen deprivation therapy, but their disease will inevitably progress to metastatic castration-resistant prostate cancer (mCRPC). Treatment failure and poor progression-free survival could be explained by the fact that PCa metastases in the same patient may be polyclonal, showing opposite responses to systemic therapies.

This project aims to recruit 100 patients with mCRPC in order to determine the prevalence of intrapatient intermetastasis polyclonality and NED using PET/CT triple-tracer PSMA/FDG/OCTREOTATE imaging and eligibility for either PSMA or OCTREOTATE radioligand therapy (RLT).

DETAILED DESCRIPTION:
Introduction: Prostate cancer (PCa) is the most common solid organ cancer in North American men. Patients becoming refractory to loco-regional therapy receive androgen deprivation therapy, but their disease will inevitably progress to metastatic castration-resistant prostate cancer (mCRPC). Of the five treatments approved for mCRPC patients, none has been shown to increase median overall survival beyond 4.8 months. Treatment failure and poor progression-free survival could be explained by the fact that PCa metastases in the same patient may be polyclonal, showing opposite responses to systemic therapies. Indeed, neuroendocrine differentiation from adenocarcinoma is often reported in metastatic PCa, which is associated with increased disease aggressiveness. Currently, no molecular tools are available to follow non-invasively mCRPC transdifferentiation and diagnose patients with neuroendocrine and/or polyclonal PCa. Positron emission tomography (PET) is a promising type of imaging using radio-labeled tracers to specifically identify tumour cells.

Hypothesis: The hypothesis of the 3TMPO clinical study is that the prevalence of intrapatient intermetastasis polyclonality can be diagnosed by combining 18F-FDG to other specific PET tracers that have the ability to non-invasively differentiate CRPC adenocarcinoma (CRPC-Adeno) (68Ga-PSMA) from neuroendocrine CRPC (CRPC-NE) tumours (68Ga-OCTREOTATE).

Objectives: The study objectives are to determine, in mCRPC patients, the prevalence of intrapatient intermetastasis polyclonality and NED using PET/CT triple tracer PSMA/FDG/OCTREOTATE imaging and their eligibility for radioligand therapy (RLT).

Method: This multicentre observational clinical study, for which prevalence of intrapatient intermetastasis polyclonality was set as the primary outcome, will recruit 100 mCRPC patients at 5 different sites across the province of Québec. 68Ga-PSMA and 18F-FDG PET scans will be performed on all enrolled patients, while 68Ga-OCTREOTATE will be performed on those presenting at least one PSMA-negative/FDG-positive lesion. The uptake of each individual lesion will be assessed for each PET tracer and patients with lesions presenting discordant uptake profiles will be considered as having polyclonal disease. OCTREOTATE-positivity will confirm the presence of CRPC-NE. PSMA or OCTREOTATE positivity of all lesions (or at least those with FDG uptake) will determine the eligibility for PSMA and OCTREOTATE RLT, respectively.

Relevance: Paradigm-shifting diagnostic and therapeutic strategies are urgently needed to improve the survival of patients with PCa and to deepen our understanding of mCRPC progression.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥ 18 years old
2. Histologically or cytologically proven PCa with or without neuroendocrine differentiation at initial diagnosis
3. Castration-resistant prostate cancer with serum testosterone ≤ 50 ng/dL (1.73 nM) anytime while on androgen deprivation therapy
4. Evidence of disease progression on prior therapy or watchful waiting. Disease progression is defined by meeting at least one of the following criteria:

   1. PSA progression defined by a minimum of 2 consecutive rising PSA levels with an interval of ≥1 week between each assessment where the PSA value at screening should be ≥1ng/ml.
   2. Soft tissue disease ONLY progression* defined by RECIST 1.1: 1) at least 20% increase in the diameter of target lesions and 2) an absolute increase of ≥ 5 mm of the sum.
   3. Soft tissue disease ONLY progression* defined as the appearance of at least one new lesion (soft tissue).
   4. Bone disease ONLY progression* defined by two or more new lesions on bone scan.
5. Metastatic disease documented by at least 3 active lesions on whole body bone scan and/or measurable soft tissue on CT-scan (lymph nodes and visceral lesions). Metastatic lesions on imaging are defined by RECIST 1.1, either:

   * ≥ 10 mm on CT scan or caliper (for lymph nodes, see below)
   * ≥ 20 mm on chest X-ray
   * lymph node ≥ 15 mm or ≥ 10 mm and having grown by ≥ 5 mm from baseline CT
   * any metastasis described on bone scan counts as a lesion
6. Able and willing to provide signed informed consent in French or English and to comply with protocol requirements.

Exclusion Criteria:

1. Another non-cutaneous malignancy or melanoma diagnosed in the past 5 years;
2. Currently under a randomized-controlled trial with unknown allocation;
3. Limited survival prognosis (ECOG ≥3);
4. Patients under dialysis;
5. Any disease or condition limiting the patient's capacity to execute the study procedures, based on the investigators' opinion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients will be enrolled in five tertiary hospital centers (CIUSSSE-CHUS, CHUQc-UL, CHUM, CIUSSS-COMTL, and MUHC) of the province of Quebec
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of INTRAPATIENT INTERMETASTATIC HETEROGENEITY | Baseline
  A patient with at least two lesions with discordant FDG/PSMA/OCTREOTATE multi-tracer imaging phenotypes.
Proportion of neuroendocrine lesion | Baseline
  Neuroendocrine lesion DEFINITION: A patient with at least one OCTREOTATE-positive lesion or histopathological features of neuroendocrine differentiation
Proportion of eligible patients for PSMA-RLT or OCTREOTATE-RLT | Baseline
  Eligibility for PSMA RLT is defined as : Having (1) at least one lesion that is PSMA-positive, and (2) no lesion that is PSMA-negative and FDG-positive. Eligibility for Octreotate RLT: Having (1) at least one lesion that is Octreotate-positive, and (2) no lesion that is Octreotate-negative and FDG-positive.

SECONDARY OUTCOMES:
18F-FDG, 68Ga-PSMA and 68Ga-OCTREOTATE positive lesions | Baseline
  POSITIVE LESION: 18F-FDG, 68Ga-PSMA and 68Ga-OCTREOTATE lesion uptake will be defined as positive if greater than that of the liver [18,19]. Using quantitative imaging methods, standardized uptake value ratio (SUVR, i.e. the ratio between lesion uptake (SUVpeak) over liver uptake (SUVmean)) will be obtained for each lesion with each tracer. For a given tracer, lesion positivity is defined as a SUVR equal or superior to 1.5.
histologic NED status of lesions | Baseline
  positive histology to synaptophysin
Pain score | Baseline and 3-months post-enrolment
  Using a Brief Pain Index (BPI) questionnaire. The severity can be expressed through 4 aspects: worst, least, average and now. The pain interference with daily activities can be represented with 7 aspects: general activity, walking, work, mood, enjoyment of life, relationships and sleep.
Physical function | Baseline and 3-months post-enrolment
  Using EQ5D questionnaire which use a 5-scale and evaluates 5 aspects: mobility, selfcare, activity, pain, anxiety and global self-evaluation.
Disease-associated symptoms | Baseline and 3-months post-enrolment
  using FACT-P questionnaire: with subscale specific for wellbeing on physical, social/family, emotional functional and prostate aspects.
PET-tracer uptake derived parameters | Baseline
  such as SUVmax, SUV mean, sum of SUVmax

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Guérin, Ph.D, Principal Investigator — Department of Nuclear Medicine,Université de Sherbrooke
Locations (5):
- Canada (5):
  - CHUM, Université de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CIUSSS du Centre-Ouest-de -l'île-de-Montreal (CIUSSS-COMTL), Montreal, Quebec
  - CHU de Québec - Université Laval (CRCHUQc-UL),, Québec, Quebec
  - Centre de recherche du CHUS (CRCHUS), Division of Urology, CIUSSS de l'Estrie - CHUS (CIUSSSE-CHUS), Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zamanian A, Rousseau E, Buteau FA, Arsenault F, Beaulieu A, April G, Juneau D, Plouznikoff N, Turcotte EE, Allard C, Richard PO, Saad F, Guerin B, Pouliot F, Beauregard JM. The tumour sink effect on 68Ga-PSMA-PET/CT in metastatic castration-resistant prostate cancer and its implications for PSMA-RPT: a sub-analysis of the 3TMPO study. Cancer Imaging. 2025 Jul 15;25(1):91. doi: 10.1186/s40644-025-00910-z. PMID 40665456